CLINICAL TRIAL: NCT07100782
Title: Estradiol-mediated Inflammation and Central Sensitization in the Pathophysiology of Endometriosis-associated Pelvic Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sawsan As-Sanie, Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00229564; R01HD108253 (NIH)
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: Relugolix Combination Therapy; Endo-EPIC (Alternative study acronym/title)
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: All investigators will be blinded to wide-spread pain (WSP) status until final analysis.
Masking Description: blind to pain
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Relugolix CT (Experimental): All participants will have the same intervention, but approximately half of those enrolled will have widespread pain and half will not.
  Approximately 65 participants with widespread pain will receive relugolix CT (relugolix 40mg, estradiol 1 mg, norethindrone acetate 0.5 mg once daily) daily for 24 weeks, and 65 participants without widespread pain will receive relugolix CT for 24 weeks.
  Interventions: Drug: Relugolix CT

INTERVENTIONS:
Drug: Relugolix CT — Study medication will be provided by Sumitomo in pill bottles containing an 84-day supply of relugolix 40mg, estradiol 1mg, norethindrone acetate 0.5mg (Relugolix Combination therapy).
  Other Names: Myfembree

SUMMARY:
The purpose of this study is to better understand how hormone suppression with Relugolix Combination-Therapy (CT) affects pelvic pain, inflammation, and pain sensitivity in women with moderate-to-severe endometriosis associated pelvic pain.

DETAILED DESCRIPTION:
All clinical activities will be performed at University of Michigan (note that recruitment may occur at locations outside of University of Michigan, such as Trinity Health, Ann Arbor, MI and Henry Ford, Detroit, MI and via social media). Endometrial biopsies will be sent via overnight courier to Dr. Jie Yu's laboratory at The University of Buffalo for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal woman between age 21 and 49 years (inclusive) at the time of consent. Menopause is defined as amenorrhea >1 year unrelated to hormonal suppression.
* History of endometriosis diagnosed by surgery (visual or biopsy confirmed), ultrasound, or MRI within 5 years of study entry
* History of self-reported moderate to severe pelvic pain for ≥ 6 months' duration at time of screening visit. Moderate-to-severe pelvic pain will be defined as self-report recall of average non-menstrual pelvic pain score over past 6 months as ≥ 4 on a 0-10 numeric rating scale (NRS)
* Willingness to participate in a relugolix CT drug intervention trial
* No use of adjunctive pain medications or on stable chronic daily use of adjunctive pain medications (excluding opioids);
* Has not used an injectable hormone therapy in the past 6 months (e.g. DepoProvera®, DepoLupron®).
* Willingness to 30-60 day washout interval of oral, vaginal, transdermal, intrauterine hormonal therapies prior to study initiation if applicable
* Willingness to use 2 forms of non-hormonal contraception during the entire duration of the study period or has had a history of a bilateral tubal occlusion procedure at least 3 months prior to screening (tubal ligation or hysteroscopic occlusion method)
* Willing to undergo quantitative sensory testing (QST), fMRI and other study procedures
* Ability to read and speak English to allow for written informed consent, phenotyping, and patient-reported outcomes measures
* Meet criteria to participate in QST and fMRI. These include:
* Normal visual acuity or correctable (with corrective lenses- glasses or contacts) to at least 20/40 for reading instructions in the MRI and visual sensitivity testing
* No contraindications to MRI (e.g., metal implants, claustrophobia)
* Willingness to refrain from pain medications such as NSAIDs, acetaminophen, and opioids for 12 hours prior to neuroimaging and QST
* Willingness to refrain from alcohol and nicotine on day of QST and neuroimaging (alcohol and nicotine consumption is allowed after testing is completed)
* Willingness to refrain from physical activity or exercise that would cause muscle and/or joint soreness for 48 hours prior to testing (routine exercise or activity that does not lead to soreness is acceptable)
* Able to lie still on their back for 1 hour during MRI

Exclusion Criteria:

* Contraindication to the use of relugolix CT (high risk of arterial or venous thrombotic, or thromboembolic disorder, known osteoporosis, current or history of breast cancer or other hormone sensitive malignancy, known hepatic impairment or disease, undiagnosed abnormal uterine bleeding, known hypersensitivity to components of relugolix CT).
* Concurrent participation in other therapeutic trials
* Pregnant, lactating, less than 6 months postpartum, or planning a pregnancy within next 12 months
* Planning pelvic or abdominal surgery during study period
* Prior major surgery in the past 4 months that involves incisions on the abdomen, chest, head, other than a skin biopsy (hysteroscopy, endometrial biopsy is ok to include).
* Planning to initiate a new adjunctive pain treatment during study treatment (e.g. cognitive behavioral therapy, physical therapy, acupuncture). Participants may be enrolled if these treatments are completed prior to trial.
* History of hysterectomy and/or bilateral oophorectomy
* Clinically significant gynecologic condition such as significant endometrial pathology (e.g. endometrial hyperplasia), persistent ovarian cyst larger than 5 cm, single fibroid 4cm or larger, more than 4 fibroids at least 2cm, or symptomatic submucosal fibroid of any size. Patients may be enrolled in this study if they were previously successfully treated for these conditions. Patients must have undergone pelvic ultrasound or MRI in the past 6 months, and provide results (or release of records to obtain results)
* History or current clinical diagnosis of vulvodynia.
* History or current evidence of psychosis, current suicide risk or attempt within 2 years of study (note: participants with mood disorders such as depression or anxiety will not be excluded)
* Chronic opioid, alcohol, and/or illicit drug use
* History of substance abuse within past one year
* Unable or unwilling to discontinue opioids analgesics within 48 hours of the dense phenotyping study visits
* Medical conditions that may significantly interfere with relugolix CT efficacy, ability to fully comply or would make it unsafe for participants to take part in the study, including but not limited to: morbid obesity with Body Mass Index > 45, uncontrolled autoimmune/inflammatory diseases, significant cardiopulmonary disease (e.g., angina, congestive heart failure, uncontrolled hypertension, severe cardiac valvular disease, Chronic Obstructive Pulmonary Disease (COPD), chronic asthma), renal or liver disease (e.g. cirrhosis, hepatitis), uncontrolled endocrine or allergic disorders (e.g., hypothyroidism, diabetes, allergic rhinitis), neurologic conditions (e.g., multiple sclerosis, prior stroke, neurological tumor), severe physical impairment (e.g., blindness, deafness, paraplegia); and active malignancy (any malignancy except for localized dermatologic cancer).
* Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigator would prevent safe or satisfactory completion of the study protocol.
* Individuals receiving or applying for compensation or disability and other aspects associated with potential secondary gain per self-report;
* Additional exclusion that prevent participation in QST and fMRI:

  1. Severe claustrophobia precluding MRI and evoked pain testing during scanning;
  2. Diagnosed peripheral neuropathy
  3. Diagnosed or self-reported epilepsy
  4. Diagnosed or self-reported visual-evoked migraines

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change score in lipopolysaccharide (LPS)-stimulated Macrophage inflammatory protein-1 alpha (MIP1-α) levels | baseline and week 12 visit
  LPS-stimulated MIP1-α levels measured from whole blood
Change score for functional magnetic resonance imaging (fMRI) connectivity of the somatosensory cortices to the default-mode network | baseline and week 12 visit
  Assessed using a functional connectivity MRI (fcMRI) at rest and applied pain

SECONDARY OUTCOMES:
Change scores for pelvic pain interference | baseline and week 12 visit
  Pain interference assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) 29+2 Profile v2.1 pain interference domain. Each domain ranges in score from 4-20 and the higher the score indicates greater pain interference in the past 7 days.
Change score for temporal summation at the forearm | baseline and week 12 visit
  Temporal summation is calculated as the mean difference in pain ratings evoked by the single stimuli and the trains of stimuli using a 0-100 NRS.

CONTACTS AND LOCATIONS:
Overall Officials: Sawsan As-Sanie, MD, MPH, Principal Investigator — University of Michigan; Andrew Schrepf, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets including participant self-report data will be uploaded into a NIH compliant data repository (NIMH Data Archive and National Institute of Child Health and Human Development (NICHD) DASH)
Supporting Information: Study Protocol, ICF
Time Frame: De-identified datasets will be made available after publication of the primary study results and/or at the conclusion of the NICHD-funded grant study period, barring any no-cost extension. Data will remain available for at least 3 years beyond the end date of the study.
Access Criteria: Data will be made publicly available through the NIH data repositories, per NIH policies including data use agreements and protection of identifying information.